CLINICAL TRIAL: NCT06280989
Title: Effect of Kinesio Taping Versus Myofascial Release on Menstrual Low Back Pain in Young Females
Brief Title: Effect of Kinesio Taping Versus Myofascial Release on Menstrual Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hala Mohamed Ahmed Morsy, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004768
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Low Back Pain
Keywords: kinesio taping; myofascial release technique
MeSH Terms: conditions — Low Back Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: kinesio taping and myofascial release technique
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- kinesio taping (Experimental): Each female will be treated by Kinesio tape which will be applied for three days (from the first day to the end of the third day of menstrual cycle) throughout 3 consecutive cycles.
  Interventions: Other: kinesio taping
- myofascial release technique (Experimental): Each female will be treated by myofascial relaxation technique which will be started at the third or fourth day of menstruation and continued till the onset of the next menstruation, 40 minutes, 3 times / week for 12 sessions through 3 consecutive menstrual cycle
  Interventions: Other: myofascial release technique

INTERVENTIONS:
Other: kinesio taping — Before treatment, all female participants will undergo an allergic test on the anterior surface of the elbow.
  To ensure cleanliness, alcohol will be used to clean the areas to be evaluated before applying the tape. The H technique will be employed to apply KT over the lumbar region. Participants will be instructed to bend forwards from the waist, and two vertical strips will be applied. These strips will stretch the Golgi tendon organ on both sides of the spine from the top of the buttock cleft upwards to a mid-point, with less than 25% stretch .
  Additionally, a horizontal strip will be attached across the left and right sacroiliac joints. This strip will be stretched to 50% of its maximum capacity,.
  Arms: kinesio taping
Other: myofascial release technique — myofascial release technique will be applied from prone on lumbar paravertebral muscles by using the olecranon of the physical therapist for 3 minutes, thoracolumbar fascia by using cross-handed hold, with hands placed on the T12-L1 levels and on the sacrum for 5 minutes without repetition and quadratus lumborum by using elbow with low pressure obliquely towards the center of the column for 7 min.
  Additionally, from supine on psoas muscle by transversal sliding of the psoas fascia. The therapist will place the hands laterally 3 cm from the umbilicus.
  Arms: myofascial release technique

SUMMARY:
the aim of this study is to investigate the efficacy of kinesio taping versus myofascial release technique on menstrual low back pain in young females

DETAILED DESCRIPTION:
: Menstrual low back pain is a prevalent condition among women. Menstrual low back pain occurrence is affected by hormonal changes. Menstrual low back pain incidence more than 40% to 50% during the menstrual phase (days 1-6) of the menstrual cycle, while the range of prevalence was 45 to 95%. It has a high prevalence among females, especially females aged 20 to 25 years old. Hormonal changes might play an important role in the formation of Menstrual low back pain and is the main cause of feeling of pain during menstrual cycle. kinesio taping and myofascial release technique play an important role in the treatment of Menstrual low back pain. this trial has two groups; one will receive kinesio taping three days and the second will receive myofascial release technique for12 sessions through 3 consecutive menstrual cycle

ELIGIBILITY:
Inclusion Criteria:

1. Healthy young virgin females suffering from menstrual low back pain diagnosed by the gynecologist.
2. Their ages will be ranged from 18-25 years' old
3. Their body mass index will be ranged from 20-25 kg/m2.
4. All females have regular menstruation
5. Their pain intensity is scored as > 4 on VAS just before or during the first 3 days of the menstruation

   -

Exclusion Criteria:

Females will be excluded from the study if they have:

1. Any orthopedic problems such as trauma at lower spine, congenital malformation at spine and scoliosis.
2. Any gynecological problem such as irregular menstrual cycle, secondary dysmenorrhea due to endometriosis, ovarian cyst, uterine fibroid and congenital malformation or pelvic inflammation.
3. Athletic females
4. Allergy to kinesio taping.

   -

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — this study for girls suffering from menstrual LBP clinically diagnosed by the gynecologist.
Enrollment: 44 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
pain intensity | up to four weeks]
  The scale that will be used the VAS ;each subject will instructed to put point on line from no pain to tolerable pain
pain pressure threshold | up to four weeks]
  will be measured by pressure algometer

SECONDARY OUTCOMES:
severity of dysmenorrhea | up to four weeks]
  will be measured by WaLIDD scale(intensity /Wong-Baker, work ability , days of pain and location). Where (0) without dysmenorrhea, (1-4) mild dysmenorrhea, (5-7) moderate dysmenorrhea, (8-12) sever dysmenorrh
Assess the function disability level | up to four weeks]
  will be assess by Oswestry Disability Index (ODI).

CONTACTS AND LOCATIONS:
Overall Officials: Manal El El shafei, lecture, Principal Investigator — Cairo University
Locations (1):
- Hala mohamed ahmed morsy, Giza, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No